CLINICAL TRIAL: NCT00889525
Title: Study of Cabergoline in Treatment of Corticotroph Pituitary Tumor
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Seth Gordhandas Sunderdas Medical College (Other)
Responsible Party: Dr Nalini S Shah, Seth Gordhandas Sunderdas Medical College& KEM Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC/104/2005
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2009-04-29 (Estimated); Status verified 2009-04

CONDITIONS: Cushing's Disease; Corticotroph Adenoma
Keywords: Cabergoline
MeSH Terms: conditions — Pituitary ACTH Hypersecretion; ACTH-Secreting Pituitary Adenoma | interventions — Cabergoline

ARMS (1):
- Cabergoline (Experimental)
  Interventions: Drug: Cabergoline

INTERVENTIONS:
Drug: Cabergoline — Dose 1 mg/week in divided doses, increased by 1 mg/week every month, to the maximum of 5 mg/week. If response is seen than the dose at which response is seen is continued until the end of the study.

SUMMARY:
This study was designed to check the efficacy of a new oral medical drug treatment, namely Cabergoline, for the treatment of Cushing Disease due to pituitary adenoma.

Background: Cabergoline is a Dopamine 2 receptor agonist. Corticotroph adenoma has shown to have the D2 receptor in in vitro studies.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Cushing's disease uncured biochemically after pituitary surgery with adenoma on histopathology

Exclusion Criteria:

* Patient's intolerance to drug or known sensitivity to ergot derivatives
* Pregnancy, lactation or female wishing to be pregnant
* Any serious medical illness
* Patient on any drugs known to have an interaction with cabergoline including antihypertensives like reserpine and methyl dopa, neuroleptics, metoclopramide, etc

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2007-11

PRIMARY OUTCOMES:
Response in term of mid night cortisol < 5.0 mcg/dl and/or Standard two day dexamethasone suppression test < 1.8 mcg/dl

CONTACTS AND LOCATIONS:
Overall Officials: Nalini S Shah, DM, Principal Investigator — Seth GSMC and KEM hospital, Mumbai
Locations (1):
- Seth GSMC & KEM hospital, Mumbai, Maharashtra, India